CLINICAL TRIAL: NCT02767986
Title: Where Culture Meets Genetics: Exploring Latinas' Causal Attributions of Breast and Colon Cancer and Mental Models of Disease Inheritance
Brief Title: Where Culture Meets Genetics: Exploring Latinas Causal Attributions of Breast and Colon Cancer and Models of Disease Inheritance
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916106; 16-HG-N106
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Colon Cancer; Breast Cancer
Keywords: Cultural Consensus; Natural History
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spanish-speaking Latinas: Women who speak Spanish as their primary language

SUMMARY:
Background:

Culture can affect the way a person thinks about illness. This can affect how they seek help for illness. It can also affect how they choose a treatment and follow it. This can lead to health disparities among certain groups of people. Breast and colon cancers are the most common cancers for Latinos. Even though they get these cancers at lower rates than other population groups, Latinos are more likely to be diagnosed with these cancers at advanced stages. Researchers want to study what Latina women immigrants believe causes breast and colon cancer and other factors they think play a role in disease. This understanding could lead to better interactions between Latinos and their doctors.

Objective:

To learn more about what Latina immigrants believe causes breast and colon cancer and other factors they think play a role in disease.

Eligibility:

Women ages 18 and older who:

Were born in Latin America

Speak Spanish

Have never had breast, ovarian, or colon cancer

Design:

Participants will be interviewed in person or over the phone. This will take up to an hour. The interview will be recorded. Participants will answer questions about:

Their family s cancer history

What they think causes breast and colon cancer

What they think plays a role in disease

...

DETAILED DESCRIPTION:
Research to understand the sources of health disparities has acknowledged that in addition to biomedical risk factors, culture plays an important role in differential health outcomes. Consequently, understanding cultural differences that may influence health behavior is key in working towards reducing these disparities. Causal attributions are a key component of individuals illness perceptions and thus impact health behaviors, which may present as health disparities at a population level. While research has explored non-Hispanic White women s causal attributions of breast cancer, less is known about Latina s beliefs about the causes of breast cancer, and little is known about causal attributions of colon cancer in any population. Understanding Latina s causal attributions of breast and colon cancer may provide insight into the determinants of cancer disparities in this population. Because a subset of both breast and colon cancers result from single gene mutations, which confer an increased risk of developing such cancers, understanding causal attributions in Latina populations is relevant to the field of genetics. This is especially true since Latinas have historically underutilized cancer genetic risk assessment counseling and testing services. As these services become a standard part of general healthcare provision, it will become increasingly important to understand ways in which different cultural groups interact with genetic information. One way this can be done is through investigating culturally informed mental models of disease risk and inheritance. This study seeks to describe causal attributions of breast and colon cancer and to explore mental models of disease inheritance among Latina immigrants . A qualitative exploratory design including interviews comprised of free-listing, ranking, and open-ended questions will be used. Participants will be recruited through the NIH Clinical Research Volunteer Program as well as using other resources within the Office of Participant Recruitment and from among individuals enrolled on other NIH Clinical Center protocols. First, we will describe Latina s causal attributions for these cancers. Next, we will use cultural consensus theory (CCT) to identify and describe common cultural models of causes of these cancers. Finally, we will explore Latina s mental models of disease inheritance using both free-listing and open-ended questions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Are a woman, 18 years of age or older
* Have immigrated to the United States from Latin America
* Speak Spanish
* Are able to meet in-person in the metro Washington, DC area

Puedes reunir los requisitos si:

* Eres mujer y tienes 18 a(SqrRoot) os de edad o m(SqrRoot)(Degree)s
* Has emigrado a los Estados Unidos desde Latinoam(SqrRoot)(Copyright)rica
* Hablas el espa(SqrRoot) ol con fluidez
* Puedes asistir en persona en la zona metropolitana de Washington, DC

EXCLUSION CRITERIA:

-NIH medical and research staff

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who speak spanish as their primary language; living in the metropolitan Baltimore/Washington, DC region
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
mental models of inheritance | baseline
  qualitative descriptions of women's understanding/thoughts about inheritance
causal attributions of colon cancer | baseline
  participants' free-lists of colon cancer causes
causal attributions of breast cancer | baseline
  participants' free-lists of breast cancer causes

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erby, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No